CLINICAL TRIAL: NCT01837680
Title: Insulin Detemir Versus Insulin NPH: A Randomized Prospective Study Comparing Glycemic Control in Pregnant Women With Diabetes
Brief Title: Glycemic Control Using Insulin Levemir Versus Insulin NPH for Diabetes in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-166
Record Dates: First submitted 2013-04-04; First posted 2013-04-23 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Diabetes, Gestational; Diabetes, Type 2
Keywords: Insulin, Long-Acting
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Insulin; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levemir (Active Comparator): Initial daily total insulin doses will be determined as per a weight based protocol depending on what trimester the patient is in. Sixty percent of the total daily insulin dose will be allotted to the morning total dose of insulin, while the remaining 40% will be allotted to the evening total dose. Of the morning dose, 2/3 will be allotted to the long acting insulin and 1/3 to short acting insulin. She will take half of the short-acting dose with breakfast and the other half with lunch. The evening insulin dose (40% of the total dose) will be divided in two: half the dose will be taken as short-acting insulin with dinner, and the other half as long acting insulin at bedtime. Doses are rounded down if decimals are present.
  Interventions: Drug: Insulin
- NPH (Active Comparator): Initial daily total insulin doses will be determined as per a weight based protocol depending on what trimester the patient is in. Sixty percent of the total daily insulin dose will be allotted to the morning total dose of insulin, while the remaining 40% will be allotted to the evening total dose. Of the morning dose, 2/3 will be allotted to the long acting insulin and 1/3 to short acting insulin. She will get the entire dose of short-acting insulin with breakfast. The evening insulin dose (40% of the total dose) will be divided in two: half the dose will be taken as short-acting insulin with dinner, and the other half as long acting insulin at bedtime. Doses are rounded down if decimals are present.
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin
  Other Names: Insulin NPH; Insulin Levemir

SUMMARY:
The aim of this study is to compare glycemic control in pregnant women treated with insulin Detemir and pregnant women treated with NPH insulin. These women are diagnosed with gestational diabetes (GDM) in the current pregnancy or have a preexisting diagnosis of type 2 diabetes (T2DM) at the onset of pregnancy. Our hypothesis is that there is no difference between these two treatment modalities in terms of glycemic control in diabetes.

DETAILED DESCRIPTION:
The experimental method will be a randomized controlled trial performed at Roosevelt Hospital in our Diabetes in Pregnancy Program (DIPP). Perinatologists managing the patient in DIPP determine when patients need further treatment with medical therapy. Patients undergoing care at DIPP may require medical intervention in the following clinical scenarios: failure of diet alone to control glycemic indices and grossly abnormal glucose tolerance screening test results suggesting disease of such severity that diet alone would not be sufficient. After verbally counseling the patient, she will be recruited for the study by the investigators. An extensive explanation of the objectives of the study will be presented to the patient, as well as written copies of the protocol and consent. After informed consent is given, patients will be randomized to management with either insulin NPH or detemir together with rapid acting insulin aspart (Novolog) with meals, as necessary. The primary outcome will be level of glycemic control defined as overall mean blood glucose in pregnancy. This is a well established measure of overall glycemic control that has been used in numerous publications in the obstetric literature on diabetes in pregnancy. Participants will be followed until they deliver, with an expected range of 6-16 weeks depending on when the patient was enrolled in the study. The mean glucose will be determined by the sum of average glucose at each visit divided by the number of visits).

ELIGIBILITY:
Inclusion criteria:

* All pregnant women with a viable singleton or multiple gestation at ≤34 weeks with gestational diabetes diagnosed in their current pregnancy requiring medical therapy. "Early diagnosis" GDM patients will also be included; which is defined as a diagnosis made prior to 24 weeks.
* Women with known preexisting type 2 diabetes that are in need of medical therapy.

Exclusion criteria:

* Patients <18 years of age
* a diagnosis of GDM outside of the gestational age stated above
* known allergy/prior adverse reaction to insulin NPH or insulin detemir.
* type 1 diabetes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States

REFERENCES:
- [Derived] Herrera KM, Rosenn BM, Foroutan J, Bimson BE, Al Ibraheemi Z, Moshier EL, Brustman LE. Randomized controlled trial of insulin detemir versus NPH for the treatment of pregnant women with diabetes. Am J Obstet Gynecol. 2015 Sep;213(3):426.e1-7. doi: 10.1016/j.ajog.2015.06.010. Epub 2015 Jun 9. PMID 26070699

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women with gestational diabetes mellitus (GDM) and type 2 diabetes mellitus (T2DM) who entered the Diabetes in Pregnancy Program were recruited from March 2013 through October 2014
Groups:
- Insulin NPH: Insulin neutral protamine Hagedorn (NPH) - Current weight was obtained at the visit and initial daily total insulin dose was determined based on patient weight (in kilograms) and trimester. In the first trimester, patient weight was multiplied by 0.7, in the second trimester by 0.8, and in the third trimester by 0.9 for the total daily dose of insulin (in units). Of the total daily insulin dose, 60% was allotted to the morning total dose of insulin, while the remaining 40% allotted to the evening total dose.
- Levemir: Insulin detemir (IDet) - Current weight was obtained at the visit and initial daily total insulin dose was determined based on patient weight (in kilograms) and trimester. In the first trimester, patient weight was multiplied by 0.7, in the second trimester by 0.8, and in the third trimester by 0.9 for the total daily dose of insulin (in units). Of the total daily insulin dose, 60% was allotted to the morning total dose of insulin, while the remaining 40% allotted to the evening total dose.
Period: Overall Study
Arm/Group | Insulin NPH | Levemir
Started | 52 | 53
Completed | 42 | 45
Not Completed | 10 | 8
Not completed — Lost to Follow-up | 2 | 2
Not completed — lack of insurance | 0 | 2
Not completed — allergic reaction | 6 | 0
Not completed — switched to oral hypoglycemic or diet | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Insulin NPH: Insulin neutral protamine Hagedorn
- Levemir: Insulin detemir (IDet)
- Total: Total of all reporting groups
Arm/Group | Insulin NPH | Levemir | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Continuous [Mean (Full Range); unit: years] | 35 [31 to 38] | 35 [32 to 38] | 35 [31 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 45 | 87
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 17 | 28
  Black | 7 | 5 | 12
  Hispanic | 12 | 15 | 27
  Native American/Alaskan | 12 | 6 | 18
  Biracial/Multiracial | 0 | 0 | 0
  Other | 0 | 2 | 2
T2DM [Count of Participants; unit: Participants] — Type 2 Diabetes Mellitus
  Participants | 7 | 7 | 14
GDM in previous pregnancies [Count of Participants; unit: Participants] | 8 | 9 | 17
Multiple gestation [Count of Participants; unit: Participants] | 2 | 3 | 5
Polycystic ovary syndrome [Count of Participants; unit: Participants] | 5 | 12 | 17
Chronic hypertension [Count of Participants; unit: Participants] | 5 | 6 | 11
Renal disease [Count of Participants; unit: Participants] | 1 | 5 | 6
Thyroid disease [Count of Participants; unit: Participants] | 6 | 8 | 14
Prepregnancy body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 28.3 [24.9 to 33.8] | 28.6 [24.4 to 31.1] | 28.4 [24.5 to 32.3]
Prepregnancy body status [Count of Participants; unit: Participants]
  Normal | 11 | 14 | 25
  Obese | 14 | 12 | 26
  Overweight | 12 | 16 | 28
  Morbidly obese | 4 | 3 | 7
Gestational age diagnosed [Median (Inter-Quartile Range); unit: weeks] | 26.1 [24.8 to 27.1] | 26.6 [25.4 to 28.2] | 26.3 [25.2 to 27.4]
Previous management [Count of Participants; unit: Participants]
  Diet | 35 | 39 | 74
  Diet, Metformin | 0 | 1 | 1
  Glyburide | 3 | 2 | 5
  Metformin | 3 | 2 | 5
  Metformin and glyburide | 1 | 0 | 1
  Other type of insulin | 0 | 1 | 1
Gestational age at entry to DIPP [Median (Inter-Quartile Range); unit: weeks] | 27.3 [23.3 to 28.5] | 28.1 [25.1 to 29.3] | 27.5 [24.1 to 29]
Gestational age insulin started [Median (Inter-Quartile Range); unit: weeks] | 29.6 [27.5 to 31.4] | 30.0 [25.1 to 31.5] | 30.0 [27.3 to 31.4]
Time between visits [Median (Inter-Quartile Range); unit: weeks] | 1.5 [1.3 to 2.0] | 1.5 [1.3 to 1.8] | 1.5 [1.3 to 1.9]

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control
Description: Overall mean glucose value of pregnancy. This will be determined by the sum of average glucose value at each visit, divided by the number of visits.
Time Frame: up to 41 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
mg/dL | 109.5 (10.0) | 107.4 (7.1)

2. Secondary Outcome: Number of Patients Obtaining Glycemic Control
Description: Number of each group that obtains glycemic control, defined as mean glucose <100mg/dl.
Time Frame: up to 41 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
Participants | 28 | 35

3. Secondary Outcome: Time to Achieve Glycemic Control
Description: Time (weeks) to achieve glycemic control, as defined as mean glucose <100mg/dl
Time Frame: up to 41 weeks
Measure: Median (Full Range); unit: weeks
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
weeks | 5 [3 to 9] | 5 [4 to 7]

4. Secondary Outcome: Average Fasting Glucose
Description: Mean fasting blood glucose in pregnancy, as determined by the sum of the mean fasting glucose at each visit divided by the number of visits
Time Frame: up to 41 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
mg/dL | 100.7 (10.1) | 97.3 (7.4)

5. Secondary Outcome: Post-prandial Blood Glucose
Description: Mean post-prandial blood glucose in pregnancy, as defined as the sum of the average post-prandial blood glucose at each visit divided by the number of visits.
Time Frame: up to 41 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
mg/dL | 115.2 (10.2) | 112.9 (8.9)

6. Secondary Outcome: Weight Gain
Description: Total weight gain in pregnancy
Time Frame: Number of pounds gained at each visit up to 41 weeks
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
lbs | 27.7 (15.3) | 28.6 (11.6)

7. Secondary Outcome: Neonatal Weight
Description: Neonatal weight was estimated for occurrence of neonatal macrosomia (≥4000g birth weight) and neonatal LGA(large for gestational age)(birth weight >90th percentile for gestational age
Time Frame: At delivery, up to 41 weeks
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
g | 3230 [2860 to 3530] | 3235 [2670 to 3620]

8. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age at delivery
Time Frame: at delivery, up to 41 weeks
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
weeks | 38.9 [37.6 to 39.3] | 38.8 [38.1 to 39.1]

9. Secondary Outcome: Maternal Hypoglycemia
Description: Number of participants with incidence of maternal hypoglycemia (<60mg/dl)
Time Frame: at delivery, up to 41 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
Participants | 11 | 16

10. Secondary Outcome: Neonatal Bilirubin
Description: Percentage of neonatal hyperbilirubinemia - data not collected
Time Frame: at birth, up to 41 weeks
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Intensive Care Admissions
Description: Number of participants with incidence of neonatal intensive care unit admissions
Time Frame: at birth, up to 41 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
Participants | 3 | 6

12. Secondary Outcome: Delivery Mode
Description: method of delivery including cesarean section, vaginal delivery, or assisted vaginal delivery - data not collected
Time Frame: at birth, up to 41 weeks
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Birth Rate
Description: Number of live birth rate
Time Frame: at birth, up to 41 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
Participants | 42 | 45

14. Secondary Outcome: Shoulder Dystocia
Description: Incidence of shoulder dystocia - data not collected
Time Frame: at birth, up to 41 weeks
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Polyhydramnios
Description: Incidence of polyhydramnios (defined as amniotic fluid index (AFI)>20 or deepest vertical pocket ≥8) - data not collected
Time Frame: at each visit in pregnancy up to 41 weeks
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Neonatal Hypoglycemia
Description: Number of participants with incidence of blood sugar <40mg/dl in neonate
Time Frame: at birth, up to 41 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin NPH | Levemir
Number analyzed (Participants) | 42 | 45
Participants | 0 | 2

ADVERSE EVENTS:
Arm/Group | Insulin NPH | Levemir
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/53
Other Adverse Events (participants affected / at risk) | 27/52 | 45/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin NPH (N=52) | Levemir (N=53)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Symptomatic hypoglycemia (Metabolism and nutrition disorders) | 11 (28) | 16 (102)
biochemical event of hypoglycemia (Metabolism and nutrition disorders) | 14 (26) | 27 (136) — glucose <60mg/dL regardless of presence or absence of symptoms
Symptomatic nocturnal event (Metabolism and nutrition disorders) | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes